CLINICAL TRIAL: NCT01188707
Title: A Clinical Phase I / II Trial of Belinostat in Combination With Erlotinib in Patients With Non-small Cell Lung Cancer
Brief Title: A Trial of Belinostat in Combination With Erlotinib in Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Dose over MTD reached
Sponsor: Herlev Hospital (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Bispebjerg Hospital (Other); Valerio Therapeutics (Industry); Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Anders Mellemgaard, MD, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU0928
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; Belinostat; Erlotinib; HDAC inhibitor; Phase I/II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — belinostat; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belinostat, Erlotinib, NSCLC (Experimental)
  Interventions: Drug: Belinostat and Erlotinib

INTERVENTIONS:
Drug: Belinostat and Erlotinib — The design of the first phase is a 3 +3 phase I trial. The Belinostat dose will start at 500 mg and will be increased with 250 mg until a maximum dose of 1500 mg, administered daily in 2/3 weeks. Each patient will at the same time receive 150 mg of Erlotinib daily continously.
  When the patient is enrolled at one dose level, there will be no further dose escalation for that individual patient.
  3 patients will be treated at each dose level.
  Other Names: Tarceva

SUMMARY:
The Belinostat-Erlotinib trial is designed as an open, non randomized phase I / II trial to assess the efficacy and safety of Belinostat in combination with Erlotinib in patients with non-small cell lung cancer who are eligible for treatment with erlotinib.

DETAILED DESCRIPTION:
Belinostat, developed by CuraGen, belongs to a new class of hydroxymat-type histone deacetylase (HDAC) inhibitors. HDAC inhibitors, including Belinostat, has shown marked in vitro and in vivo activity against a number of solid tumors and hematological cancers. Belinostat has proven to be effective as a single agent or in combination with other anticancer agents such as doxorubcin, paclitaxel, carboplatin, fluorouracil, bortezumib, and there has been observed synergy between Belinostat or other HDAC inhibitors and EGFR inhibitors gefinitinib and erlonitib.

Furthermore, the antineoplastic activity of Belinostat seen in preclinical experiments have resulted in only moderate toxicity.

In the two Phase I trials of Belinostat for solid tumors and hematological malignancies Belinostat have been well tolerated at doses up to 2000 mg daily in more than 100 patients.

Fatigue, nausea and vomiting has been the main side effects and with none or very mild hematologic toxicity. Approximately 25% of patients in the study of solid tumors achieved stable disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent of an approved informed consent form
2. A. For the dose escalation phase: Patients with histological or cytological confirmed non-small cell lung cancer who are rated suitable for treatment with Erlotinib B. For MTD expansion phase: Patients diagnosed with non- small cell lung cancer rated suitable for treatment with Erlotinib and with measurable disease according to RECIST version 1.1
3. Performance status (ECOG) ≤ 2
4. Life expectancy at least 3 months
5. Age ≥ 18 years
6. Acceptable liver, kidney and bone marrow function, defined as:

   * Bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * ASAT, ALAT and alkaline phosphatase ≤ 3 x ULN (if liver metastases is ≤ 5 x ULN allowed)
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
   * WBC> 2.5 x 109 / l, neutrophils> 1.0 x 109 / l, platelets> 100 x 109 / l
   * Hemoglobin> 9.0 g / dl or> 5.6 mmol / l
7. Acceptable coagulation: PT and APTT within ≤ 1.5 x ULN or in the therapeutic range if given anticoagulant
8. A negative pregnancy test for women of childbearing age. In fertile men and women the use of effective contraception methods are required during the trial
9. Serum potassium within normal range

Exclusion Criteria:

1. Treatment with experimental drugs within the last 4 weeks
2. Former anti-cancer therapy within the last 3 weeks before the start of experimental treatment, including chemotherapy, radiotherapy, endocrine therapy or immunotherapy
3. Simultaneous presence of active infection or other concomitant present medical condition likely to affect the experimental procedures, including significant cardiovascular disease (New York Heart Association Class III or IV heart disease, myocardial infarction within the past 6 months, unstable angina, congestive heart failure requiring treatment, unstable arrhythmia or the need for antiarrhythmic drugs or signs of ischemia on ECG, marked baseline prolongation of QT / QTc interval, for example repeated demonstration of a QTc interval> 500 msec; long QT syndrome; required the use of concurrent medication on dosage belinostat days, which may cause torsades de pointes (see Appendix 1).
4. Altered mental status that prevents understanding of the informed consent process and / or execution of the necessary experiments
5. Secondary malignancy present (previous malignancy accepted if cured by treatment for > 3 years ago)
6. Intestinal obstruction or threatening bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  The primary purpose of the phase I part of the trial is to establish the tolerance dose (maximum tolerated dose (MTD) and dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Efficacy | 1 year
  The phase II part of the study is to assess the efficacy of Belinostat and Erlotinib in combination assessed by disease control rate, defined as non - progression at 3 months / Stable disease or better) using RECIST response criteria version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jon L Andersen, MD, Principal Investigator — Dept of Oncology Copenhagen University Hospital Herlev
Locations (1):
- Dept of Oncology Copenhagen University Hospital Herlev, Copenhagen, Denmark